## "Tolerance to Baked Foods in Children Under 6 Years Old Allergic to Cow's Milk and Egg Proteins"

PIC-104-14

## **INFORMED CONSENT FORM**

| I,, parent/legal guard, have read and understood the s | |
|---|---|
| any questions I had, and they have been clearly answered. | stady information. Thave asked |
| I voluntarily consent forto unde challenge to baked cow's milk/egg, conducted in the Allergy Uni | |
| Signature of Parent/Guardian: Name: ID: | |
| Signature of Child (if over 12 years old): Name: | |
| Signature of Informing Physician: Name: | |
| Esplugues, date: | |